CLINICAL TRIAL: NCT02833792
Title: A Phase IIa Study of Allogeneic Human Mesenchymal Stem Cells in Subjects With Mild to Moderate Dementia Due to Alzheimer's Disease
Brief Title: Allogeneic Human Mesenchymal Stem Cells for Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stemedica Cell Technologies, Inc. (Industry)
Collaborators: Stemedica International SA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STEM105-M-AD
Record Dates: First submitted 2016-06-20; First posted 2016-07-14 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cells (Experimental): Stem cells
  Interventions: Drug: Human Mesenchymal Stem Cells and Lactated Riunger's Solution
- Placebo (Placebo Comparator): Lactated Ringer's Solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Human Mesenchymal Stem Cells and Lactated Riunger's Solution — Intravenous administration
  Arms: Stem Cells
Other: Placebo — Intravenous administration
  Arms: Placebo

SUMMARY:
STUDY OBJECTIVES

Primary:

To assess the safety and tolerability of ischemia-tolerant allogeneic human mesenchymal stem cells (hMSCs) manufactured by Stemedica versus placebo administered intravenously to subjects with mild to moderate dementia due to Alzheimer's disease.

Secondary:

To assess the preliminary efficacy of hMSCs versus placebo in subjects with Alzheimer's-related dementia, as evidenced by neurologic, functional, and psychiatric endpoints.

DETAILED DESCRIPTION:
This is a Phase IIa multi-center, randomized, single-blind, placebo-controlled, crossover study in subjects with mild to moderate dementia due to Alzheimer's disease. Only the subject and their caregiver will be blinded to the study treatment. The study will consist of two cohorts of subjects (20 subjects per cohort), randomized in a 1:1 allocation to receive active study drug or placebo. Cohort 1 will receive a single intravenous dose of hMSCs of 1.5 million cells per kilogram body weight on their Study Day 1, and Cohort 2 will receive equal volume of Lactated Ringer's Solution on their Study Day 1. At the six-month time point for each subject after their first infusion, Cohort 1 will receive a single intravenous dose of Lactated Ringer's Solution and Cohort 2 will receive a single intravenous dose of hMSCs at 1.5 million cells per kilogram of the subject's body weight. Approximately 40 subjects will be enrolled in this study. An independent Data and Safety Monitoring Board will conduct periodic safety reviews.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 55-80 years of age.
2. Diagnosed with mild to moderate dementia for at least 3 months prior to enrollment, based on the National Institute of Neurological and Communicative
3. Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINDS-ADRDA) Alzheimer's criteria.
4. MMSE between 12-24 (inclusive) at time of enrollment.
5. Amyloid-positive florbetapir PET scan.

Exclusion Criteria:

1. Prior treatment with stem cells.
2. History of intracranial, subdural, or subarachnoid hemorrhage.
3. Subjects with baseline brain MRI showing more than four (4) cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), and/or one (1) or more areas of superficial siderosis, and/or evidence of a prior macrohemorrhage. MRI must include fluid-attenuation inversion recovery (FLAIR) and T2*-weighted gradient-recalled-echo (GRE) sequences.
4. History of cancer within the past 5 years, with the exception of localized basal or squamous cell carcinoma.
5. History of seizure disorder.
6. Diagnosis of cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL).
7. History of cerebral neoplasm.
8. Myocardial infarction within six months of enrollment.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of aMBMC administration | 18 months
  Number of patients with adverse events will be reported

SECONDARY OUTCOMES:
Efficacy of aMBMC administration | 18 months
  Changes is scores relatively to baseline using NIHSS system will be reported for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Lev Verkh, PhD, Study Chair — Stemedica Cell Technologies
Locations (1):
- John Wayne Cancer Institute @ Providence St. John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor information — http://stemedica.com